CLINICAL TRIAL: NCT06449222
Title: A Phase II, Multi-site, Randomized, Open-label Clinical Trial to Evaluate the Safety, Efficacy, and Pharmacokinetics of BNT327 at Two Dose Levels in Combination With Chemotherapeutic Agents as First- and Second-line Treatment in Triple-negative Breast Cancer
Brief Title: Safety and Preliminary Effectiveness of BNT327, an Investigational Therapy for Breast Cancer, When Given in Combination With Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT327-02
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Breast Cancer; Triple Negative Breast Cancer; Metastatic Triple Negative Breast Cancers
Keywords: Programmed Death-1; Programmed Death Ligand-1; Programmed Death-1 monoclonal antibodies; Anti vascular endothelial growth factor-A (anti-VEGF-A)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Carboplatin; Gemcitabine; Paclitaxel; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 Arm 1 - BNT327 DL1 + Nab-paclitaxel (Experimental)
  Interventions: Drug: BNT327 Dose Level 1 (DL1); Drug: Nab-placlitaxel
- Cohort 1 Arm 2 - BNT327 DL2 + Nab-paclitaxel (Experimental)
  Interventions: Drug: BNT327 Dose Level 1 (DL2); Drug: Nab-placlitaxel
- Cohort 2 Arm 1 - BNT327 Optimized dose + Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel; Drug: BNT327 Optimized Dose
- Cohort 2 Arm 2 - BNT327 Equivalent Q3W dose + Gemcitabine + Carboplatin (Experimental)
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: BNT327 Equivalent Q3W Dose
- Cohort 2 Arm 3 - BNT327 Equivalent Q3W dose + Eribulin (Experimental)
  Interventions: Drug: Eribulin; Drug: BNT327 Equivalent Q3W Dose

INTERVENTIONS:
Drug: BNT327 Dose Level 1 (DL1) — Intravenous (IV) infusion
  Arms: Cohort 1 Arm 1 - BNT327 DL1 + Nab-paclitaxel
Drug: BNT327 Dose Level 1 (DL2) — IV infusion
  Arms: Cohort 1 Arm 2 - BNT327 DL2 + Nab-paclitaxel
Drug: Nab-placlitaxel — IV infusion
  Arms: Cohort 1 Arm 1 - BNT327 DL1 + Nab-paclitaxel; Cohort 1 Arm 2 - BNT327 DL2 + Nab-paclitaxel
Drug: Carboplatin — IV infusion
  Arms: Cohort 2 Arm 2 - BNT327 Equivalent Q3W dose + Gemcitabine + Carboplatin
Drug: Gemcitabine — IV infusion
  Arms: Cohort 2 Arm 2 - BNT327 Equivalent Q3W dose + Gemcitabine + Carboplatin
Drug: Paclitaxel — IV infusion
  Arms: Cohort 2 Arm 1 - BNT327 Optimized dose + Paclitaxel
Drug: Eribulin — IV infusion
  Arms: Cohort 2 Arm 3 - BNT327 Equivalent Q3W dose + Eribulin
Drug: BNT327 Optimized Dose — IV infusion
  Arms: Cohort 2 Arm 1 - BNT327 Optimized dose + Paclitaxel
Drug: BNT327 Equivalent Q3W Dose — IV infusion
  Arms: Cohort 2 Arm 2 - BNT327 Equivalent Q3W dose + Gemcitabine + Carboplatin; Cohort 2 Arm 3 - BNT327 Equivalent Q3W dose + Eribulin

SUMMARY:
This study is a Phase II, multi-site, randomized, open-label clinical study to evaluate the safety, efficacy, and pharmacokinetics (PK) of BNT327 at two dose levels in combination with chemotherapeutic agents in the first- and second-line treatment of participants with locally advanced/metastatic triple-negative breast cancer (mTNBC).

DETAILED DESCRIPTION:
Participants will be treated until disease progression, intolerable toxicity, participant withdrawal, death, study termination or up to 2 years (whichever occurs first).

The study plans to randomize or assign eligible participants into two cohorts, i.e., Cohort 1 and Cohort 2. In Cohort 1, participants will be randomized to two treatment arms investigating two dose levels of BNT327 in combination with Nab-paclitaxel. Participants in Cohort 2 will be assigned to one of three treatment arms by their clinician.

Cohort 2 will not begin until the appropriate dose to move forward has been determined from Cohort 1. After this, the arms in Cohort 2 exploring different chemotherapy combinations will begin to enroll.

Participants in Cohort 2, Arm 1 will receive the optimal dose of BNT327 in combination with paclitaxel. Participants in Cohort 2, Arms 2 and 3, will receive the equivalent dose of BNT327 administered once every 3 weeks (Q3W) in combination with gemcitabine plus carboplatin (Arm 2), or eribulin (Arm 3).

ELIGIBILITY:
Inclusion Criteria:

* Have given informed consent by signing and dating an informed consent form before initiation of any study-specific procedures.
* Male or female, aged ≥18 years at the time of giving informed consent.
* Are willing and able to comply with scheduled visits, the treatment schedule, the planned study assessments (including participant completed diaries) and other requirements of the study. This includes that they are able to understand and follow study-related instructions.
* Have confirmed locally recurrent inoperable or mTNBC as defined by the most recent American Society of Clinical Oncology (ASCO) / College of American Pathologists (CAP) guidelines. Note, participants initially diagnosed with hormone receptor-positive and/or HER2-positive breast cancer must have histological confirmation of TNBC in a tumor biopsy obtained from a local recurrence or distant metastasis site.

  * Systemic treatment naïve locally advanced/metastatic participants are eligible if:

    * They have received no prior systemic therapy in the locally advanced unresectable/metastatic setting including chemotherapy, immunotherapy, or investigational agents.
    * They have completed treatment for Stage I-III breast cancer, if indicated, and ≥6 months has elapsed between the completion of treatment with curative intent (e.g., date of primary breast tumor surgery or date of last adjuvant chemotherapy administration, or date of last radiation therapy, whichever occurred last) and first documented local or distant disease recurrence. This also includes participants initially diagnosed with hormone receptor-positive and/or HER2-positive breast cancer prior to TNBC diagnosis.
  * Participants who received one prior systemic therapy in the locally advanced/metastatic setting are eligible if:

    * They have received one systemic chemotherapy in the metastatic setting and have progressed on first line therapy. Radiographic progression must have been documented. Radiographic progression is defined as unequivocal progression of existing tumor lesions or developing new tumor lesions as assessed by the investigator.
    * They have had a recurrence-free interval of ≥6 months if they have received treatment with curative intent in the past. A recurrence-free interval of ≥6 months is required for all participants (both first- and second-line treatment settings) who have received prior treatment for breast cancer with curative intent.
* Have provided a tissue sample, archival or fresh, during the screening period (bone biopsies, fine needle aspiration biopsies, and samples from pleural or peritoneal fluid are not acceptable; participants with only one target lesion are not eligible to provide a biopsy). If an archival tumor sample is not available, the participant must undergo a fresh biopsy, if medically feasible to be eligible for the study.
* Have at least one measurable lesion as the targeted lesion based on RECIST version 1.1. Lesions treated after prior local treatment (radiotherapy, ablation, interventional procedures) are generally not considered as target lesions. If the lesion with prior local treatment is the only targeted lesion, evidence-based radiology must be provided to demonstrate disease progression (the single bone metastasis or the single central nervous system metastasis should not be considered as a measurable lesion).
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Have a minimum life expectancy of >3 months.
* Have adequate organ function, as defined below:

  * Hematology:

    * Absolute neutrophil count ≥1.5 × 10^9/L (without G-CSF support within two weeks prior to Cycle 1, Day 1).
    * Platelet count ≥100 × 10^9/L (without transfusion within 2 weeks prior to Cycle 1, Day 1).
    * Hemoglobin ≥90 g/L or 5.6 mmol/L. Note: Criterion must be met without packed red blood cell transfusion or without erythropoietin dependency within the prior 2 weeks before receiving the first dose of study treatment.
  * Liver function:

    * Total bilirubin ≤1.5 × upper limit of normal (ULN).
    * With Gilbert's syndrome total bilirubin <3 mg/dL and direct bilirubin ≤ULN. Note, Gilbert's syndrome must be documented appropriately as past medical history.
    * Participants without liver metastasis alanine aminotransferase and aspartate aminotransferase ≤2 × ULN.
    * Participants with liver metastasis alanine aminotransferase and aspartate aminotransferase ≤5 × ULN.
    * Albumin ≥3.0 g/dL.
  * Renal function: Creatinine clearance ≥50 mL/min. Cockcroft-Gault formula. Note, in participants who will be treated with gemcitabine plus carboplatin, creatinine clearance should be ≥60 mL/min.
  * Qualitative urine protein ≤1+. If qualitative urine protein ≥2+, a 24-hour urine protein quantitative test is required. If the 24-hour urine protein result is <1 g, the participant can be enrolled.
  * Coagulation function: International normalized ratio or prothrombin time and activated partial thromboplastin time ≤1.5 × ULN unless the participant is receiving anticoagulation therapy as long as prothrombin or activated partial thromboplastin is within therapeutic range of intended use of anticoagulant.
* Are women of childbearing potential (WOCBP) who have a negative serum beta human chorionic gonadotropin pregnancy test. Women who are postmenopausal (defined as 12 months with no menses without an alternative medical cause) or permanently sterilized (verified by medical records) will not be considered WOCBP and therefore will not be required to undergo pregnancy testing.
* Are WOCBP who agree to practice a highly effective form of contraception and to require the use of barrier contraception methods, starting at at the time of giving informed consent and continuously until 6 months after receiving the last study treatment.
* Are men who are sterile or if they are potentially fertile (i.e., are not surgically [e.g., have had a vasectomy] or congenitally sterile) and sexually active with a partner of childbearing potential, who agree to use condoms and to ask their sexual partners to practice a highly effective form of contraception during the study, starting at the time of giving informed consent and continuously until 6 months after receiving the last dose of IMP.
* Agree not to donate germ (ova, oocytes, sperm) for the purposes of assisted reproduction during study, starting at the time of giving informed consent and continuously until 6 months after receiving the last dose of IMP.

Exclusion Criteria:

* Are pregnant or breastfeeding or are planning pregnancy or planning to father children during the study or within 6 months after the last dose of IMP.
* Have a medical, psychological, or social condition which, in the opinion of the investigator, could compromise their wellbeing if they participate in the study, or that could prevent, limit, or confound the protocol-specified assessments or procedures, or that could impact adherence to protocol described requirements.
* Have received any of the following therapies or drugs prior to the initiation of study:

  * Participants who received prior treatment with a PD(L)-1/Vascular Endothelial Growth Factor bispecific antibody.
  * Have received a systemic anticancer regimen within 4 weeks prior to the initiation of study treatment or have received palliative radiotherapy within 7 days prior to the initiation of study treatment, or have received any other chemotherapy, curative/palliative radiotherapy, biologic therapy (including tumor vaccines, cytokines, or growth factors for tumor control) or any experimental antitumor drugs within 4 weeks prior to the initiation of study treatment.
  * Have received other systemic immunostimulatory agents or immunosuppressive therapies (such as interferon-alpha [IFN-α], interleukin-2 [IL-2], or methotrexate) within 4 weeks prior to the initiation of study treatment or are within five half-lives of the treatment drug (whichever is longer). Exception: Excluding local, intranasal, intraocular, intra-articular or inhaled corticosteroids, short-term use (≤7 days) of corticosteroids for prophylaxis (e.g., prevention of contrast agent allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity reactions caused by exposure to allergens).
  * Have received systemic corticosteroids (at a dosage greater than 10 mg/day of prednisone or an equivalent dose of other corticosteroids) within 3 weeks prior to the initiation of study treatment.
  * Have been vaccinated with live attenuated vaccine(s) within 4 weeks prior to initiation of study treatment.
  * Received broad-spectrum IV antibiotics therapy within 3 weeks prior to initiation of study treatment.
  * Use of any non-study investigational medicinal product within five half-lives of first dose or within 4 weeks, whichever is longer, before initiation of study treatment in this study or ongoing participation in the active treatment phase of another interventional clinical study.
* Have undergone major organ surgery (core needle biopsies are allowed >7 days prior study start), significant trauma, or invasive dental procedures (such as dental implants) within 28 days prior to the initiation of study treatment or plan to undergo elective surgery during the study. Placement of vascular infusion devices is allowed.
* Have received allogeneic hematopoietic stem cell transplantation or organ transplantation.
* Have spinal cord compression or central nervous system metastases that is untreated and symptomatic or requires treatment with corticosteroids or anticonvulsants for associated-symptom control. Exception: Treated brain metastases which is no longer symptomatic and for which no corticosteroid or anticonvulsant treatment is needed (the participant must be recovered from the acute toxic effect of radiotherapy; study treatment assignment must be ≥2 weeks after completion of radiotherapy).
* Have active autoimmune disease that has required systemic treatment in the past 2 years (e.g., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Those who had a history of autoimmune diseases with anticipated relapse (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for those with clinically stable autoimmune thyroid disease or type 1 diabetes.
* Have had other malignant tumors within 2 years prior to the study treatment are not allowed. Except for those: who have been cured with local treatment (such as basal cell or squamous cell carcinoma of the skin, superficial or non-invasive bladder cancer, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, and papillary carcinoma of thyroid; including prostate cancer with CR within the past 3 years).
* Have any of the following heart conditions within 6 months prior to the study treatment:

  * Acute coronary syndrome, coronary artery bypass grafting, congestive heart failure, aortic dissection, stroke, or other Grade 3 and above cardiovascular and cerebrovascular events.
  * New York Heart Association functional classification ≥II heart failure or left ventricular ejection fraction <50%.
  * Those who have ventricular arrhythmias requiring clinical intervention, second- to third-degree atrioventricular block, or congenital long QT syndrome. Participants with treated cardiac arrythmia/atrial fibrillation are allowed.
  * Mean QT interval corrected by Fridericia's method (QTcF) >480 ms (the ECG can be repeated at the discretion of the investigator).
  * Use of cardiac pacemaker.
  * Cardiac troponin I or T >2 x ULN.
* Have any of the following hypertension or diabetic conditions prior to initiation of study treatment:

  * Poorly controlled diabetes (fasting blood glucose ≥13.3 mmol/L [240 mg/dL] or HbA1C [≥8.5%]).
  * Uncontrolled hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥90 mmHg) while on antihypertensive medicine.
  * A history of hypertensive crisis or hypertensive encephalopathy.
* Have serious non-healing wounds, ulcers, or bone fractures. This includes history of abdominal fistula, tracheoesophageal fistula, gastrointestinal perforation, or intra abdominal abscess for which an interval of 6 months must pass before the Screening Visit. In addition, the participant must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing the fistula/perforation.
* Participants with evidence of major coagulation disorders or other significant risks of hemorrhage such as:

  * History of intracranial hemorrhage or intraspinal hemorrhage.
  * Tumor lesions invading large blood vessels and are at significant risk of bleeding.
  * Had clinically significant hemoptysis or tumor hemorrhage of any cause within 1 month prior to the initiation of study treatment.
* Have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Participants with indwelling catheters (e.g., PleurX) are allowed.
* Have uncontrolled tumor-related pain requiring analgesic treatment not managed by a stable analgesic regimen. For asymptomatic metastatic lesion, if its growth may cause dysfunction or intractable pain (e.g., current epidural metastasis unrelated to spinal cord compression), local treatment should be considered before screening, if appropriate.
* Have a known or suspected hypersensitivity to the study treatments including any active ingredient or excipients thereof.
* Have a known human immunodeficiency virus infection or known acquired immunodeficiency syndrome, with the following exceptions:

  * Participants with cluster of differentiation 4 (CD4)+ T-cell (CD4+) counts ≥350 cells/µL per local laboratory should generally be eligible for the study.
  * Participants who have not had an opportunistic infection within the past 12 months.
* Have a known history/positive serology for hepatitis B requiring active antiviral therapy (unless immune due to vaccination or resolved natural infection or unless passive immunization due to immunoglobulin therapy). Individuals with positive serology must have hepatitis B virus viral load below the limit of quantification.
* Have active hepatitis C virus infection; individuals who have completed curative antiviral treatment with hepatitis C virus viral load below the limit of quantification are allowed.
* Are subject to exclusion periods from another investigational study.
* Are vulnerable individuals, i.e., are individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. This includes all sponsor, study site, or third party (e.g., CRO, vendor) personnel directly involved in the conduct of the study and their family members or dependents, as well as all study site personnel otherwise supervised by the investigator.
* Participants with AEs from prior antitumor therapy that have not returned to Grade 1 (graded by NCI CTCAE version 5.0 criteria) or below (unless the investigator determines that certain AEs pose no safety risk to participants, such as hair loss, Grade 2 peripheral neuropathy or stable hypothyroidism under hormone replacement therapy) are not eligible for the study.
* Have superior vena cava syndrome or symptoms of spinal cord compression.
* Those with active, or a history of, pneumonitis requiring treatment with steroids, or has active, or a history of, interstitial lung disease. Those with a history of pulmonary fibrosis, or currently diagnosed with severe lung diseases such as interstitial pneumonia, pneumoconiosis, chemical pneumonitis, or any other condition resulting in significant impairment in lung function. Exception: Asymptomatic interstitial changes caused by previous radiation therapy, chemotherapy, or other factors such as smoking are acceptable.
* Have active tuberculosis or history of tuberculosis that was not successfully treated.
* Have underlying condition(s) that may increase risk of the combination treatment or complicate the interpretation of toxicities and AEs, as judged by the investigator, or other scenarios that the investigators consider the participant is not eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events (TEAEs), adverse events of special interest (AESIs), treatment emergent serious adverse events (SAEs) | up to 100 days after the last dose of treatment
  In the combination treatment regimen according to the (US) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 (CTCAE version 5.0). By treatment arm and overall.
Occurrence of dose interruption, dose reduction, and discontinuation of study treatment due to adverse events (AEs) | up to 100 days after the last dose of treatment
  By treatment arm and overall.
Objective Response Rate (ORR) | Until end-of-treatment visit, i.e., up to 24 months after the first dose of treatment
  Defined as the proportion of participants in whom a confirmed complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1] based on the investigator's assessment) is observed as best overall response. By treatment arm.
Best percentage change from baseline in the tumor size | Until end-of-treatment visit, i.e., up to 24 months after the first dose of treatment
  Based on the investigator's tumor assessment according to RECIST 1.1. Defined as the change from baseline in percent to the minimal tumor size until tumor progression/recurrence or death (whichever occurs first). By treatment arm.
Proportion of participants who have achieved early tumor shrinkage | up to 4 months after first dose of treatment
  Defined as ≥10% decrease in the pretreatment sum of diameters at first post-treatment tumor scan in target lesions. By treatment arm.

SECONDARY OUTCOMES:
PK assessment: Maximum concentration (Cmax) derived from serum concentration of BNT327 | from pre-dose to 15 days after study treatment
  By treatment arm for Cohort 1, Arm 1 and 2, and Cohort 2, Arm 1
PK assessment: Area Under the Curve During the Dosing Interval (AUCtau) derived from serum concentration of BNT327 | from pre-dose to 15 days after study treatment
  If data permits. By treatment arm for Cohort 1, Arm 1 and 2, and Cohort 2, Arm 1
Incidence of detectable BNT327 antidrug antibodies in serum | from pre-dose to 100 days after last dose of study treatment
ORR as assessed by the investigator | Until end-of-treatment visit, i.e., up to 24 months after the first dose of treatment
  As assessed by the investigator (Cohort 2)
Duration of Response (DOR) | Until end-of-treatment visit, i.e., up to 24 months after the first dose of treatment
  Defined as the time from first objective response (CR or PR per RECIST 1.1) to first occurrence of objective tumor progression or death from any cause, whichever occurs first based on investigator's review
Disease Control Rate (DCR) | Until end-of-treatment visit, i.e., up to 24 months after the first dose of treatment
  Defined as the proportion of participants in whom a confirmed CR or PR or stable disease (per RECIST 1.1, stable disease assessed at least 6 weeks after first dose) is observed as best overall response based on the investigator's review.
Time to Response (TTR) | Until end-of-treatment visit, i.e., up to 24 months after the first dose of treatment
  Defined as the time from randomization/assignment to first objective response (CR or PR per RECIST 1.1) based on the investigator's review.
Progression-Free Survival (PFS) | up to 24 months after completion of study treatment of the last participant
  Based on investigator's review tumor assessment according to RECIST 1.1 is defined as the time from randomization/assignment to first confirmed objective tumor progression (progressive disease per RECIST 1.1), or death from any cause, whichever occurs first.
PFS rate | up to 24 months after completion of study treatment of the last participant
  As measured at 6, 12, 18, and 24 months
Overall Survival (OS) | up to 24 months after completion of study treatment of the last participant
  Defined as the time from randomization/assignment to death from any cause
OS rate | up to 24 months after completion of study treatment of the last participant
  As measured at 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (62):
- United States (30):
  - Arizona Oncology Associates, PC, Tucson, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Stanford University School of Medicine - Stanford Cancer Institute (SCI) - Stanford Women's Cancer Center, Palo Alto, California
  - Saint John's Health Center - John Wayne Cancer Institute (JWCI), Santa Monica, California
  - Rocky Mountain Cancer Centers (RMCC), Denver, Colorado
  - Yale University - Yale Cancer Center, New Haven, Connecticut
  - Hematology Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Kaiser Permanente - Moanalua Medical Center And Clinic, Honolulu, Hawaii
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Carle Foundation Hospital d/b/a Carle Cancer Center, Urbana, Illinois
  - Northwest Cancer Centers, P.C., Dyer, Indiana
  - Community Health Network, Indianapolis, Indiana
  - Helen G. Nassif Community Cancer Center, Cedar Rapids, Iowa
  - Henry Ford Hospital, Detroit, Michigan
  - HealthPartners Regions Specialty Clinics, Saint Louis Park, Minnesota
  - Minnesota Oncology - Woodbury Clinic, Woodbury, Minnesota
  - Bozeman Health Deaconess Hospital Cancer Center, Bozeman, Montana
  - Rutgers Cancer Institute of NJ (Rutgers, The State University of New Jersey), New Brunswick, New Jersey
  - Stony Brook University Hospital, Stony Brook, New York
  - Clinical Research Alliance Inc., Westbury, New York
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - The West Clinic, P.C. d/b/a West Cancer Center, Germantown, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Ut Health Science Center - San Antonio (UTHSCSA), Cancer Therapy & Research Center, San Antonio, Texas
  - Bon Secours St. Francis Medical Center, Midlothian, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington
- Australia (5):
  - Icon Cancer Care, Wesley Clinic, Auchenflower
  - Peninsula Oncology Centre, Frankston
  - Peter MacCallum Cancer Centre, Melbourne
  - Mater Hospital Sydney, Sydney
  - Westmead Hospital, Westmead
- Turkey (Türkiye) (19):
  - Baskent Universitesi Tip Fakultesi Adana Hastanesi, Adana
  - Medical Park Seyhan Hospital, Adana
  - Adana City Training and Research Hospital, Adana
  - Sakarya University - Faculty of Medicine, Adapazarı
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Hacettepe Universitesi Kanser Enstitusu, Ankara
  - Sbu Dr.A.Y. Ankara Onkoloji SUAM, Ankara
  - Memorial Ankara Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Gaziantep Sanko University Medical Faculty, Gaziantep
  - Koc Universitesi Hastanesi (Koc University Hospital), Istanbul
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istinye Universitesi Bahcesehir Liv Hospital, Istanbul
  - Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Yeditepe University Hospital, Istanbul
  - Medical Point Izmir Hospital, Izmir
  - Ondokuz Mayis Universitesi Tip Fakultesi, Samsun
  - Acibadem Adana Hospital, Seyhan
  - Gazi University Medical Faculty, Yenimahalle
- United Kingdom (8):
  - Stoke Mandeville Hospital - Buckinghamshire Healthcare NHS Trust, Aylesbury
  - Hull and East Yorkshire Hospitals NHS Trust - Castle Hill Hospital, Cottingham
  - Edinburgh Cancer Centre-Western General Hospital, Edinburgh
  - St James's University Hospital - Leeds Teaching Hospitals NHS Trust, Leeds
  - St Bartholomew's Hospital - Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Sarah Cannon Research Institute, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biteghe FAN, Mungra N, Malindi Z, Chalomie NET, Stanislas KA, Yasmin-Karim S, Mike Makrigiorgos G, Chipidza FE, Akinrinmade OA, Sridhar S, Barth S, Ngwa W. The Therapeutic Potential of Photoimmunotherapy as a Safe, Effective and Non-Toxic Treatment Option for Superficial Triple Negative Breast Cancer. Cancer Med. 2025 Sep;14(18):e71255. doi: 10.1002/cam4.71255. PMID 40970572